CLINICAL TRIAL: NCT00283790
Title: Investigation of Psycliomotor and Cognitive Residual Effects After Single Oral Doses of Zolpidem Tartrate Extended Release 12.5 mg and Eszopielone 3 mg Compared to Placebo in Healthy Young Volunteers, Using Plurazepam 30 mg As An External Comparator
Brief Title: Residual Effects of Zolpidem Tartrate Extended Release and Eszopiclone Vs Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PM_L_0289
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

INTERVENTIONS:
Drug: zolpidem tartrate

SUMMARY:
Investigation of Psychomotor and Cognitive Residual Effects of Single Oral Doses of Zolpidem Tartrate Extended Release 12.5 mg and Eszopiclone 3 mg Compared to Placebo in Healthy Young Volunteers, Using Flurazepam 30 mg as an External Comparator

DETAILED DESCRIPTION:
This is a crossover study, with 4 different treatments (Ambien, Lunesta, placebo, and flurazepam). The flurazepam arm always comes last due to the long washout period associated with it. The other 3 arms are randomized.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Healthy male and female subjects aged between 18 and 45 years.
2. Usual bedtime between 21:00 and 01:00
3. Body mass index (BMI) between 18 and 32 kg/m2.
4. Certified as healthy by a comprehensive clinical assessment (detailed medical history and a complete physical examination).
5. Laboratory tests within the normal range of the laboratory (hematology, biochemistry, urinalysis) or within the acceptable range per agreement between investigator and sponsor.
6. Negative urine pregnancy test for females (to be confirmed at screening and prior to every dose of study medication)
7. Women must use a medically acceptable form of contraception (steroidal contraceptive, double-barrier, or intra-uterine device) during the entire study period, or they must be surgically sterilized or post-menopausal. If abstinent, women must agree to use double-barrier contraception throughout the study period should they become sexually active.
8. Written informed consent signed

EXCLUSION CRITERIA:

1. Presence or history of clinically relevant cardiovascular, hepatic, pulmonary, gastrointestinal, renal, metabolic, hematological, neurologic or psychiatric disease, any acute infectious disease or signs of acute illness, and myasthenia gravis
2. Any disorder initiating or maintaining sleep such as Obstructive Sleep Apnea, Insomnia, Restless Leg Syndrome, Periodic Limb Movement Disorder, Circadian Rhythm Disorder and Parasomnia
3. Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
4. Symptomatic hypotension, whatever the decrease of blood pressure, or asymptomatic postural hypotension defined by a decrease in SBP equal to or greater than 20 mmHg within two minutes when changing from the supine to the standing position.
5. History of hypersensitivity to zolpidem, eszopiclone, or flurazepam.
6. Use of any medication within one month prior to study start, except occasional use of acetaminophen or ibuprofen.
7. History of drug abuse during prior twelve months
8. Excessive consumption of xanthine-based beverages (more than 6 cups or glasses per day) or unable to stop consumption during the overnight study periods.
9. Inability to communicate or cooperate with the investigator because of a language problem, poor mental status, or impaired cerebral status.
10. Positive results of urine drug screen testing (amphetamines, benzodiazepines, cannabis, barbiturates, cocaine, opiates, antidepressants).
11. Any use of dietary, herbal, and/or fitness/body-building supplements (with the exception of vitamins)
12. Current use of tobacco products including cigarettes, cigars, pipes, or chewing tobacco, current participation in a smoking cessation program, or discontinuation of smoking within 3 months prior to screening
13. Subject is currently participating in another clinical trial with an investigation product/device (or within 30 days of screening).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36
Dates: Start 2006-01; Study Completion 2006-04

PRIMARY OUTCOMES:
Psychometric testing:
Critical Flicker Fusion (CFF)
Choice Reaction Time (CRT)
Immediate and Delayed Recall of Supraspan Word Lists (WRI and WRD)
Compensatory Tracking Task (CTT)
Digit Symbol Substitution Test (DSST)

SECONDARY OUTCOMES:
Efficacy Measures:
Sleep measures from Morning Sleep Questionnaire
Residual Effects of Zolpidem Tartrate Extended Release and Eszopiclone Vs Placebo
Leeds Sleep Evaluation Questionnaire (LSEQ)
Bond & Lader (B&L) Visual Analog Scale
Health Outcome Measures
Sleep Treatment Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States